CLINICAL TRIAL: NCT01785095
Title: Prospective, Open-label, Uncontrolled Clinical Trial Evaluating Multiple Controlled Ovarian Hyperstimulation Cycles in Oocyte Donor, to Assess the Immunogenicity of FSH-IBSA
Brief Title: Immunogenicity of Repeated Follicle Stimulating Hormone (FSH) Stimulation Cycles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11E/FSH03
Record Dates: First submitted 2013-01-23; First posted 2013-02-07 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Oocyte Donation
MeSH Terms: interventions — Follicle Stimulating Hormone, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FSH (Experimental): FSH (Follicle stimulation hormone, 75 IU/vial) will be administered to women according to their need and response assessed by the Investigator.
  Interventions: Drug: FSH (Follicle Stimulating Hormone)

INTERVENTIONS:
Drug: FSH (Follicle Stimulating Hormone)

SUMMARY:
The purpose of the study is to evaluate immunogenic potential of FSH-IBSA in healthy volunteers undergoing controlled ovarian hyperstimulation (COH) in an oocyte donation program.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers undergoing controlled ovarian hyperstimulation for oocyte donation with the following characteristics:
* Able and willing to sign the Subject Consent Form and adhere to the study visit schedule;
* >=18 and <35 years old;
* Regular menstrual cycle (26 - 35 days);
* BMI between 18 and 30 kg/m2;
* First gonadotrophin treatment (i.e. naïve Subjects with regard to exposure to human derived or recombinant gonadotrophins);
* basal FSH <10 IU/L and E2 <80 pg/ml (~290 pmol/l);
* Normal TSH levels;
* Willing to perform at least two consecutive oocyte retrieval cycles (with a wash out period of two months).

Exclusion Criteria:

* Age <18 and >=35 years;
* PCOS;
* Endometriosis;
* Subjects with evidences of autoimmune or rheumatic diseases;
* Hypersensitivity to the active substance or to any of the excipients (lactose);
* Abnormal bleeding of undetermined origin;
* Subject found to be positive to anti-TSH antibodies (i.e. suffering from thyroidal diseases);
* Uncontrolled adrenal dysfunction;
* Neoplasia;
* Severe impairment of renal and/or hepatic function;
* Use of concomitant medications that might interfere with study evaluations (e.g. immunosuppressant, non-study hormonal medications, therapeutics proteins like insulin, growth hormone…).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dep.Obstet-Gynec.-Reproduction,Institut Universitari Dexeus, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Follicle Stimulation Hormone: FSH (Follicle stimulation hormone, 75 IU/vial) will be administered to women according to their need and response assessed by the Investigator.
  FSH (Follicle Stimulating Hormone)
Period: Overall Study
Arm/Group | Follicle Stimulation Hormone
Started | 27
Completed | 24
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: All the subjects that started the stimulation.
Arm/Group | Follicle Stimulating Hormone
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.7 (5.4)
Gender [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 21.7 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Producing Anti-FSH Antibodies.
Description: The immunogenicity potential of FSH in healthy volunteer will be assessed by analysing serum samples collected at different timepoints during two treatment cycle for oocytes donation: cycle 1, serum samples will be collected before treatment start (baseline), after 7-13 days and after 28 days of treatment; Cycle 2: serum samples will be collected before starting the second cycle (baseline 2), after 7-13 days and after 28 days of treatment. Cycle 1 and cycle 2 will be separated by a wash-out period of two months.
Time Frame: 4 months.
Population: presence of Antibodies against FSH
Measure: Number; unit: participants
Arm/Group | Follicle Stimulationg Hormone
Number analyzed (Participants) | 27
participants | 0

2. Secondary Outcome: Number of Oocytes Retrieved
Description: the number of oocytes retrieved in the first cycle and in the second cycle are compared.
Time Frame: after 2 weeks of treatment
Measure: Mean (Standard Deviation); unit: oocytes
Groups:
- First Cycle: First treatment cycle.
- Second Cycle: Second treatment cycle performed after 1 month of wash out.
Arm/Group | First Cycle | Second Cycle
Number analyzed (Participants) | 27 | 24
oocytes | 13.4 (7.7) | 15.7 (7.8)

3. Secondary Outcome: Total Dose of FSH Units Used.
Time Frame: after 2 weeks of treatment
Measure: Mean (Standard Deviation); unit: IU
Groups:
- Second Cycle: Second treatment cycle after 1 month of wash out.
Arm/Group | First Cycle | Second Cycle
Number analyzed (Participants) | 27 | 24
IU | 1911.1 (604.8) | 1984.4 (622.4)

ADVERSE EVENTS:
Arm/Group | Follicle Stimulating Hormone
Serious Adverse Events (participants affected / at risk) | 1/27
Other Adverse Events (participants affected / at risk) | 7/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Follicle Stimulating Hormone (N=27)
Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) — post oocyte retrieval haemorrhage
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Follicle Stimulating Hormone (N=27)
abdominal pain (Gastrointestinal disorders) | 1 (2)
Pirexia (General disorders) | 1 (1)
bacterial vaginosis (Infections and infestations) | 1 (1)
candida infection (Infections and infestations) | 1 (1)
lymp injury (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headhache (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No